CLINICAL TRIAL: NCT00786851
Title: Salvage Treatment With Lenalidomide and Dexamethaosne(LEN-DEX) in Patients With Relapsed/Refractory Mantle Cell Lymphoma (MCL)
Brief Title: Salvage Treatment With Lenalidomide and Dexamethaosne (LEN-DEX) in Patients With Relapsed/Refractory Mantle Cell Lymphoma (MCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIL LEN-DEX MCL 07; EudraCT Number 2008-000044-14
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: MANTLE CELL LYMPHOMA
Keywords: MANTLE CELL LYMPHOMA (MCL); Lenalidomide (Len); Dexamethasone (Dex)
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Lenalidomide will be supplied as 5 mg and 25 mg capsules for oral administration.Dexamethasone (Soldesam 0.2%) will be supplied as 20 mg liquid for oral administration (1 bottle = 20 mg; daily dose = 2 bottles = 40 mg).
  Interventions: Drug: Lenalidomide and Dexametasone

INTERVENTIONS:
Drug: Lenalidomide and Dexametasone — Lenalidomide will be supplied as 5 mg and 25 mg capsules for oral administration.Dexamethasone (Soldesam 0.2%) will be supplied as 20 mg liquid for oral administration (1 bottle = 20 mg; daily dose = 2 bottles = 40 mg).

SUMMARY:
This is a prospective, multicenter phase II trial designed to evaluate the safety and activity of the combination of Lenalidomide (Len) and Dexamethasone (Dex) in patients with relapsed/refractory mantle cell lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MCL
* Understand and voluntarily sign an informed consent form;
* Able to adhere to the study visit schedule and other protocol requirements;
* Age ≥ 18;
* Patients treated with at least one prior treatment regimen, not eligible for or relapsed after more intensive treatments (stem cell transplant);
* Patients with refractory or relapsed disease;
* Measurable and/or valuable disease;
* Adequate haematological counts: ANC > 1.5 x 109/L and platelet count > 75 x 109/L unless due to bone marrow involvement by MCL;
* Conjugated bilirubin up to 2 x ULN unless due to liver involvement by MCL;
* Alkaline phosphatase and transaminases up to 2 x ULN unless due to liver involvement by MCL;
* Creatinine clearance ≥ 50 ml/min;
* HIV negativity;
* HCV negativity;
* HBV negativity or patients with HBcAb +, HbsAg -, HBs Ab+/- and anti HBV prophylaxis with lamivudine;
* Non peripheral neuropathy or CNS disease;
* Life expectancy > 6 months;
* Performance status < 2 according to ECOG scale;Disease free of prior malignancies (a part MCL) with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast;
* Written informed consent;
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed;

Exclusion Criteria:

* Patients who have received an experimental drug or used an experimental medical device within 4 weeks before the planned start of treatment. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study;
* CNS disease (meningeal and/or brain involvement by lymphoma);
* TVP in the last year;
* History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances;
* Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug);
* Creatinine clearances < 50 ml/min;
* HIV positivity;
* HBV positivity with the exception of patients with HBVcAb +, HbsAg -, HBs Ab+/- in anti HBV prophilaxis with lamivudine;
* Pregnant or lactating women;
* Hypersensitivity reactions to previous thalidomide (if any);
* Prior rash ≥ 3 while taking thalidomide (if any);
* Active opportunistic infection;
* Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To explore the antitumor activity of the association of Len-Dex in term of overall (OR) and complete response (CR) in patients with relapsed/refractory MCL | 3 years

SECONDARY OUTCOMES:
To explore the safety profile; | 2 years
To explore the modification of tumoral neo-angiogenic biomarkers and the relationship with response to Len-Dex therapy; | 2 years
To evaluate the clinical efficacy of Len-Dex in terms of response duration (RD) and overall survival (OS). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, MD, Study Director — Ospedale S. Maria della Misericordia, Udine
Locations (17):
- Italy (17):
  - Ospedale SS. Antonio Biagio e Cesare Arrigo, Alessandria
  - Centro diriferimento oncologico, Aviano (PN)
  - Ematologia Spedali Civili, Brescia
  - Ematologia Ospedale Businco, Cagliari
  - Fondazione IRCCS UO Ematologia 1, Milan
  - Ospedale Niguarda Cà granda, Milan
  - Ospedale San Raffaele Ematologia, Milan
  - Università Policlinico San Matteo Divione di Ematologia, Pavia
  - AO Bianchi Melacrino Morelli UO Ematologia, Reggio Calabria
  - AO Arcispedale S.Maria Nuova Ematologia, Reggio Emilia
  - Università La Sapienza Ematologia, Roma
  - Istituto Clinica Humanitas, Rozzano (MI)
  - AO Universitaria di Sassari Istituto di Ematologia, Sassari
  - Policlinico Le Scotte Clinica Ematologica, Siena
  - Osp. San Giovanni Battista Ematologia2, Torino
  - Osp. Cardinalle Panico Divisione di Ematologia, Tricase (LE)
  - AO Universitaria clinica Ematologica ed Unità terapie Cellulari Carlo Melzi, Udine

REFERENCES:
- [Derived] Zaja F, De Luca S, Vitolo U, Orsucci L, Levis A, Salvi F, Rusconi C, Ravelli E, Tucci A, Bottelli C, Balzarotti M, Brusamolino E, Bonfichi M, Pileri SA, Sabattini E, Volpetti S, Monagheddu C, Vacca A, Ria R, Fanin R. Salvage treatment with lenalidomide and dexamethasone in relapsed/refractory mantle cell lymphoma: clinical results and effects on microenvironment and neo-angiogenic biomarkers. Haematologica. 2012 Mar;97(3):416-22. doi: 10.3324/haematol.2011.051813. Epub 2011 Nov 4. PMID 22058200